CLINICAL TRIAL: NCT00452010
Title: Pain Reducing Effect of Transcutaneous Electrical Nerve Stimulation (TENS) in Patients With Chronic Low Back Pain or Chronic Lumbo-radiculalgia and Followed in Pain Treatment Centers
Brief Title: Pain Reducing Effect of Transcutaneous Electrical Nerve Stimulation in Patients With Chronic Low Back Pain or Lumbo-radiculalgia
Acronym: LOBOTENS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Françoise LORCA, CHU de Saint-Etienne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0601001; lombotens
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Low Back Pain; Chronic Lumbo-radiculalgia
Keywords: TENS; chronic low back pain; chronic lumbo-radiculalgia; placebo; Roland scale

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): transcutaneous electrical nerve stimulation
  Interventions: Device: CEFAR PRIMO TENS Class IIA (active)
- 2 (Placebo Comparator): No transcutaneous electrical nerve stimulation
  Interventions: Device: CEFAR PRIMO TENS Class IIA (no active)

INTERVENTIONS:
Device: CEFAR PRIMO TENS Class IIA (active) — Active TENS. 4 sessions per day during 3 months.
  Arms: 1
Device: CEFAR PRIMO TENS Class IIA (no active) — Placebo TENS. 4 sessions per day during 3 months.
  Arms: 2

SUMMARY:
Prior studies showed contradictory results about the best type of TENS in chronic pain pathology.

Therefore we want to evaluate the efficacy assessment of TENS on patients with chronic low back pain or chronic lumbo-radiculalgia.

The functional ability score is evaluated by the Roland scale at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Stable chronic low back pain or stable chronic lumbo-radiculalgia
* Patients with a pain score at least superior or equal to 4
* Patients followed in pain clinics
* Written informed consent

Exclusion Criteria:

* Prior ambulatory TENS practice
* Lumbo-radiculalgia pathology surgery within 3 months before inclusion
* Acute low back pain or bilateral lumbo-radiculalgia
* Acute radiculalgia
* Surgery planned within 6 months
* Pacemaker
* Symptomatic low back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
functional ability | Week 6

SECONDARY OUTCOMES:
pain relief | Week 6 and Month 3
functional repercussions by Roland scale | Month 3
functional repercussions by Dallas scale | Month 3
quality of life | Day 1 and Month 3
global satisfaction of cares | Month 3
medical consumption | From Day 1 to Month 3
TENS observance | from Day 1 to Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Bernard LAURENT, Professor, Principal Investigator
Locations (8):
- France (8):
  - CHU d'Amiens, Amiens
  - CHU de Grenoble, Grenoble
  - CHU de Limoges, Limoges
  - Fondation Hôpital Saint Joseph - MARSEILLE, Marseille
  - La Timone - MARSEILLE, Marseille
  - Centre Catherine de Sienne - Nantes, Nantes
  - CHU de Saint-Etienne, Saint-Etienne
  - CH de Voiron, Voiron

REFERENCES:
- [Result] Buchmuller A, Navez M, Milletre-Bernardin M, Pouplin S, Presles E, Lanteri-Minet M, Tardy B, Laurent B, Camdessanche JP; Lombotens Trial Group. Value of TENS for relief of chronic low back pain with or without radicular pain. Eur J Pain. 2012 May;16(5):656-65. doi: 10.1002/j.1532-2149.2011.00061.x. Epub 2011 Dec 20. PMID 22337531